CLINICAL TRIAL: NCT05761873
Title: Comparing Paper Letters in Addition to Emailed Audit and Feedback in Refining Asthma Treatment to Improve Clinical and Environmental Results in Primary Care
Brief Title: Letters in Addition to Emailed Audit and Feedback in Refining Asthma Treatment in Primary Care
Acronym: CLEARAIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leeds (Other)
Collaborators: NHS West Yorkshire Integrated Care Board (Unknown)
Responsible Party: Principal Investigator, Owen Thomas, Principle investigator, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CLEARAIR321442
Record Dates: First submitted 2023-02-27; First posted 2023-03-09 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Asthma
Keywords: Paper; Email; Audit and Feedback; Behavioural Change Taxonomy; Inhalers; Climate change; Environment; Carbon dioxide; pMDI; DPI; Spacer; Primary care; Prescribing; Theoretical Domains Framework
MeSH Terms: conditions — Asthma | interventions — Paper

STUDY DESIGN:
Intervention Model Description: The study design is a cluster Randomised Controlled trial, where primary care practices within the NHS West Yorkshire ICB region would be randomised by Primary Care Network (PCN) to receive either paper copies of A&F reports and emailed PDF A&F reports, or emailed PDF A&F reports alone. The research team will randomise (using a simple computerised Random Number Generator) each cluster of PCN practice pseudonyms to receive their audit and feedback report either by email alone, or by email and a physical copy through the post. To prevent contamination effects and for ease of analysis, cluster randomisation would be utilised on a Primary Care Network (PCN) basis. Once randomised, each practice will receive 7 A&F reports over the course of a year in their allocated format, informing them of their progress.
Who Masked: Investigator
Masking Description: The research team will remain blinded to the identity of which practice has been assigned which pseudonym. However, clearly it is impossible for the ICB and the practices themselves to be blinded to the assignment status of each practice due to the nature of the intervention. The ICB will retain the process of sending out reports by email and post, as would be standard practice in such a quality improvement project.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paper audit and feedback only (Active Comparator): Provision of A&F reports by email (standard practice in the region) to allocated practices depending on randomisation status.
  Interventions: Other: Provision of audit and feedback via paper only
- Paper and email audit and feedback (Experimental): Provision of A&F reports by paper via the post (new intervention being trialled) and email (standard practice) to allocated practices depending on randomisation status.
  Interventions: Other: Provision of audit and feedback via email and paper

INTERVENTIONS:
Other: Provision of audit and feedback via email and paper — Provision of A&F reports by paper via the post (new intervention being trialled) and email (standard practice) to allocated practices depending on randomisation status.
  Arms: Paper and email audit and feedback
Other: Provision of audit and feedback via paper only — Provision of A&F reports by email (standard practice in the region) to allocated practices depending on randomisation status.
  Arms: Paper audit and feedback only

SUMMARY:
Public Health England have estimated that 36,000 excess deaths occur each year due to UK air pollution. Respiratory inhalers produce 3% of NHS greenhouse gas production. The two main inhaler device categories are pressurised Metered Dose Inhalers (pMDIs) and Dry Powder Inhalers (DPIs). The chemical propellant in pMDIs is the majority cause of inhaler carbon footprint, with pMDIs having an 18 times higher carbon footprint than DPIs. The rates of asthma in the UK population are amongst the highest worldwide and its mortality rate remains amongst the worst in Europe.

A pre-existing Audit and Feedback (A&F) quality improvement project (QIP) is being undertaken by NHS West Yorkshire Integrated Care Board (ICB) with the aim of improving asthma outcomes and reducing the environmental impact of inhalers in primary care. The A&F being utilised here has been validated locally in two peer reviewed studies and is now standard practice in the region. There is convincing evidence that A&F has a positive effect on enacting behaviour change, especially where behaviour change is related to prescribing with low baseline compliance with guidelines. However, the evidence base is poor on which design features of A&F produce enhanced results. There is supporting evidence from local studies suggesting that posted paper A&F may be more effective at producing behaviour change than emailed copies of A&F alone.

This study seeks to randomise the primary care practices within the pre-arranged QIP, to receive either a paper and emailed A&F report bimonthly for the duration of the study period, or to receive an emailed A&F report alone. The primary outcome of the study would be a comparison of the number of 'low-global warming potential' inhalers prescribed as a percentage of the total prescribed inhalers from each intervention group.

DETAILED DESCRIPTION:
A small collection of drug categories used by the health service produce a disproportionate amount of the total NHS greenhouse gas production, namely respiratory inhalers and anaesthetic gases (3% and 2% of total NHS production respectively). Inhalers are the mainstay of treatment for a variety of chronic respiratory conditions, offering a unique mechanism of drug delivery directly to the lungs to maximise effect and limit systemic side-effects. Four main inhaler device categories exist, including the pressurised Metered Dose Inhaler (pMDI - developed in the 1950s), the Dry Powder Inhaler (DPI - developed in the 1980s), the Breath-Actuated metered dose Inhaler (BAI), and the Soft Mist Inhaler (SMI - developed in the 2000s - currently only available to provide a long-acting muscarinic receptor antagonist). Since the 1990s, the pMDIs have been powered through hydrofluorocarbons (HFCs) - a greenhouse gas calculated to be 3800 times more powerful than that of carbon dioxide. This chemical propellant found in BAIs and pMDIs - rather than the medication itself - is the majority cause of the high carbon footprint related to all inhaler therapy, with pMDIs having an 18 times higher carbon footprint than DPIs.

There are no clear national guidelines on the clinical decision-making process of choosing between a pMDI or a DPI. To operate a DPI, there is a minimal Peak Expiratory Flow Rate (PEFR) required of between 20-50 L/min to overcome the device's internal resistance, with optimal PERF being between 40-65 L /min; this is often described as requiring a quick, deep breath creating turbulent flow to aid drug delivery (26). For a pMDI, a slow breath generating a PERF of around 30 L/min is optimal. A small study of healthy children found that while 100% of children age 5 could use a DPI with a flow rate of 30 L/min, only 62.5% could use one requiring 60 L/min; these numbers increased to 100% and 91.7% respectively for children aged 6. NICE recommended in 2000 that DPIs should be avoided for children under the age of 5. A literature review of inhaler technique studies highlighted that pMDIs require skilled coordination between actuation and inhalation for optimal drug delivery, which is not the case with DPIs. This review indicates that patients who struggle with pMDI coordination are often children and elderly patients, and they suggest that better technique is often achieved where one inhaler device type alone is used in a patient's care.

Although a pMDI may be preferred to a DPI in some clinical scenarios, England has a disproportionately high usage of pMDIs compared to its European neighbours; pMDIs were shown to make up 71.6% of all prescribed inhalers in England, compared to <50% in the rest of Europe and between 10-30% in Scandinavia (31,32). Given these figures, work has been undertaken in England to explore the effect of switching from pMDIs to DPIs in asthma. A post-hoc analysis from the Salford Lung Study (2236 patients) showed that moving to a DPI from a pMDI-based maintenance therapy more than halved their associated carbon footprint. Patients moved to DPIs also experienced consistently superior clinical outcomes compared to their baseline care and the majority of patients opted to remain on the DPI after switching. A large survey of UK asthma patients identified that 65% were unaware of the environmental impacts of pMDIs, with 60% of pMDI patients being open to switching their device type.

As previously stated, England has a significantly higher burden of disease from asthma compared with many other comparable countries, with that burden falling unequally on society in patterns determined by typical social determinants of health such as socioeconomic status. With two thirds of asthma deaths being linked to preventable factors, there is scope in this region to make significant health gains for the population whilst taking major strides to decrease health inequalities. The RCP report into asthma deaths produced a number of key recommendations for medical and professional care, signifying that all asthma patients should: be provided with a personal asthma action plan (PAAP); have a structured asthma review with an assessment of inhaler technique at least annually; be assessed for evidence of overuse of short-acting reliever and those that do should be invited for urgent review; be monitored for poor adherence to preventer inhaled corticosteroids; and be encouraged to use combination inhalers. There is notable overlay between the goals of improving asthma outcomes and improving the environmental impacts of asthma therapy, with both having a focus on using the right type of inhaler for the right patient and ensuring patients use effective inhaler techniques that optimises drug delivery whilst minimises waste.

Audit and feedback (A&F) is defined by Ivers et al. as the "provi(sion of) a recipient with a summary of their performance over a specified period of time" and has long history of use within a diverse area of research and business to promote clinician and organisational behaviour change. In healthcare, A&F has been used either alone, or as part of a composite quality improvement project (QIP), to improve health practitioner practice on the basis of guidelines or targets. A 2012 Cochrane review systematically reviewed 140 papers on A&F spanning several decades and produced a meta-analysis showing an absolute risk difference (RD) in practitioners changing behaviour to comply with preferred practice of 4.3% (interquartile range 0.5% to 16%). Their investigation emphasised that A&F is particularly effective when it is targeted specifically at prescribing practices (mean adj. RD 13.1% verses diabetes management 0.5%) and where baseline compliance is low. The authors hypothesised that this is because prescribing is a less complex behaviour that may be perceived by health practitioners as important. Meta-regression of the Cochrane data showed that the effect size of A&F has remained largely unchanged over the last two decades of study, leading the authors to postulate that there is no longer reasonable clinical equipoise to question if A&F is effective. However, they also conclude that studies aiming to isolate how A&F can be utilised most effectively by comparing different A&F variations are few and far between and that this should be the target of future A&F research. From the few studies that do exist comparing types of A&F, the meta-analysis showed that it is most effective when: a supervisor or respected colleague delivers the feedback; feedback is frequently presented; there are both specific goals and action-plans; focuses on decreasing a behaviour; there is low baseline performance; and when non-physicians are the focus of intervention.

A&F has previously been used successfully within the West Yorkshire Clinical Commissioning Group (CCG) - now replaced by the NHS West Yorkshire Integrated Care Board (ICB) - to effect change on primary care prescribing practices. The ASPIRE cluster Randomised Controlled Trial (cRCT) of A&F in this region produced a reduction in risky prescribing (odds ratio 0.82), while the CROP quasi-experimental controlled interrupted time series analysis of A&F correlated with 15,000 fewer patients being inappropriately prescribed opioids over a period of a year compared to controls. Both studies utilised a similar A&F design, utilising a theoretical structure based around the Theoretical Domains Framework (TDF) that is ideal for determining the possible perceptions of interventions by its intended targets. They also operated the Behaviour Change Taxonomy (BCT) to describe their employed behavioural change techniques along with their intended effects. A qualitative process evaluation of the CROP study identified that there was a possible preference for paper A&F copies of A&F compared to emailed PDF A&F, as it allowed for easier sharing for colleague discussion and made the report easier to 'flick' through. Some participants however preferred the emailed PDF, or to have both paper and emailed PDF, stating that it facilitated sharing in larger teams.

The American production company 'Pitney Bowes Inc' produced a report in 2008 combining open access internal reports on the greenhouse gas contribution of direct mail from a variety of global mail companies - including Royal Mail - to give an indicative range of CO2 emissions per letter between 10 to 30 grams of carbon dioxide (median of 17.9 grams per letter). It is clear there is a question on whether paper copies of A&F, in addition to emailed PDF copies, could enhance the clinician response to an intervention. If this is found to be the case, it may be that the added greenhouse gas produced from the paper A&F is considerably outweighed by the improved intervention effect in reducing the use of high global-warming potential inhalers.

As part of a pre-existing quality improvement work, the NHS West Yorkshire ICB will be initiating a year-long project of the proven A&F techniques described above to bring about prescribing behaviour change. The aim of this work will be to initiate several asthma-related prescribing behaviour changes within this primary care region, including the increased use of appropriate 'low-global warming potential' inhalers. This A&F report schedule will be based on designs previously shown within the ASPIRE and CROP studies to produce clinically and statistically significant reductions in inappropriate prescribing within this primary care locality. The report construction will be supported by the University of Leeds (UoL) primary care research team under prior agreed arrangements between NHS West Yorkshire ICB and individual practices. All non-anonymised data used to construct the final reports will be processed exclusively in-house by NHS West Yorkshire ICB. After this year long QIP, fully anonymised data - aggregated by primary care practice - will be shared with the UoL Primary Care research team under prior agreed data sharing arrangements between NHS West Yorkshire ICB and individual practices to allow the team to undertake statistical monitoring of the impacts of the QIP.

As previously stated, there is currently a knowledge gap in how A&F can be best implemented to produce the most effective behaviour change. From previous published qualitative investigation of the CROP A&F intervention, it is clear that there is equipoise around whether A&F is enhanced when provided in paper format, as opposed to a virtual format alone. Here we propose a cluster RCT to address this question, where primary care practices within the NHS West Yorkshire ICB who are already scheduled to take part in a planned A&F QIP will be randomised to either receive their A&F in a virtual email PDF format alone, or to receive both an emailed and paper format PDF report through the post. To prevent contamination effects and for ease of analysis, cluster randomisation would be utilised on a Primary Care Network (PCN) basis. To analyse the results of this study, additional required data from NHS West Yorkshire ICB would be necessary to identify which anonymised, aggregate practice datasets were randomised to which arm of the trial via the use of pseudonyms. To achieve this, the ICB will assign each practice a pseudonym before the study, and the University of Leeds research team will randomise (using a simple computerised random number generator) each pseudonym to an intervention group to receive their feedback either by email alone, or email and a physical copy in the post. This information will then be passed back to the ICB.

ELIGIBILITY:
Inclusion Criteria:

* Must be a primary care practice in the West Yorkshire ICB region.
* Must consent to data sharing, and not opted out of the West Yorkshire QIP

Exclusion Criteria:

* Not a primary care practice in the West Yorkshire ICB region.
* A primary care practice that has not consented to data sharing, or opted out of the West Yorkshire QIP

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2023-04-24 (Actual); Primary Completion 2024-05-17 (Actual); Study Completion 2025-04-17 (Actual)

PRIMARY OUTCOMES:
High-global warming potential' pMDI inhalers use | 1 year
  The number of 'high-global warming potential' preventer pMDI inhalers prescribed as a proportion of the total prescribed preventer inhalers for patients with asthma from each primary care practice - limited to those aged over 5.

SECONDARY OUTCOMES:
6 or more SABA's prescriptions | 1 year
  Total number of patients with 6 or more SABA's prescription issues per a year in the last 12 months
12 or more SABA's prescriptions | 1 year
  Total number of patients with 12 or more SABA's prescription issues per a year in the last 12 months
3 or less inhaled corticosteroids prescriptions | 1 year
  Total number of patients with 3 or less inhaled corticosteroids prescription issues in the last 12 months
2 or more courses of oral prednisolone prescriptions | 1 year
  Total number of patients with 2 or more courses of oral prednisolone prescription issues in the last 12 months?
Children with second-hand smoke status recorded | 1 year
  Percentage of patients aged between 6-19 with asthma, with second-hand smoke status recorded
Combination prescriptions of salbutamol MDIs with DPI preventers | 1 year
  Patients prescribed a combination of salbutamol MDIs with DPI preventers
Prescriptions of non-salbutamol MDI's Vs DPIs prescribed in over 12s | 1 year
  Percentage of non-salbutamol MDI's Vs DPIs prescribed in over 12s

CONTACTS AND LOCATIONS:
Overall Officials: Owen Thomas, MBBS, Principal Investigator — University of Leeds
Locations (1):
- White Rose House, Wakefield, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Overall data will be used to construct internal reports, support conference presentations, and peer reviewed scientific papers. Pseudo-anonymised IPD may be used to support a publication via a secure storage database.

REFERENCES:
- [Background] Ivers NM, Sales A, Colquhoun H, Michie S, Foy R, Francis JJ, Grimshaw JM. No more 'business as usual' with audit and feedback interventions: towards an agenda for a reinvigorated intervention. Implement Sci. 2014 Jan 17;9:14. doi: 10.1186/1748-5908-9-14. PMID 24438584
- [Background] Ivers N, Jamtvedt G, Flottorp S, Young JM, Odgaard-Jensen J, French SD, O'Brien MA, Johansen M, Grimshaw J, Oxman AD. Audit and feedback: effects on professional practice and healthcare outcomes. Cochrane Database Syst Rev. 2012 Jun 13;2012(6):CD000259. doi: 10.1002/14651858.CD000259.pub3. PMID 22696318
- [Background] Alderson SL, Farragher TM, Willis TA, Carder P, Johnson S, Foy R. The effects of an evidence- and theory-informed feedback intervention on opioid prescribing for non-cancer pain in primary care: A controlled interrupted time series analysis. PLoS Med. 2021 Oct 4;18(10):e1003796. doi: 10.1371/journal.pmed.1003796. eCollection 2021 Oct. PMID 34606504
- [Background] Wood S, Foy R, Willis TA, Carder P, Johnson S, Alderson S. General practice responses to opioid prescribing feedback: a qualitative process evaluation. Br J Gen Pract. 2021 Sep 30;71(711):e788-e796. doi: 10.3399/BJGP.2020.1117. Print 2021 Oct. PMID 33979300